CLINICAL TRIAL: NCT03571867
Title: Comparison of The Severity of Agitation of Sugammadex and Atropine-Nesostigmine in Adenotonsillectomy in Pediatric Patients? : a Double Blind Randomised Clinical Trial
Brief Title: Comparison of The Severity of Agitation of Sugammadex and Atropine-Nesostigmine in Adenotonsillectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Havva Sayhan, assistant professor, Sakarya University
Other Study IDs: sugammadex
Record Dates: First submitted 2018-06-05; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: The Severity of Agitation in Adenotonsillectomy in Pediatric Patients
Keywords: Adenotonsillectomy; Severity of Agitation; Sugammadex

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group Sugammadex: After surgery, while the TOF count was 2/4, the residual muscle relaxation was antagonized with 2 mg/kg iv sugammadex + 0.01 ml/kg saline in Group S
- group Neostigmine: After surgery, while the TOF count was 2/4, the residual muscle relaxation was antagonized with 0.02 mg/kg neostigmin+0.01 mg/kg atropine in Group N.

SUMMARY:
the use of sugammadex during the reversal of neuromuscular blocking after adenotonsillectomy surgery in pediatric patients would be advantageous in terms of patient comfort and reducing side effects. Thus, we aimed to evaluate the time to extubation, agitation and pain scores in pediatric patients who underwent adenotonsillectomy and awakened with neostigmine and sugammadex in our study.

DETAILED DESCRIPTION:
A total of 70 patients in the American Society of Anesthesiologists (ASA) I-II risk group, aged 5-13 years, who will be undergoing adenotonsillectomy with recurrent / chronic tonsillitis or obstructive sleep apnea in the otorhinolaryngology clinic of our hospital were included. Investigator did not assign specific interventions to the study participants. Patients were selected to sugammadex + saline group (Group S) and neostigmin+atropine group (Group N) and 35 patients were seleceted for each group randomly. Patients receive interventions as part of routine medical care, and a researcher studies the effect of the intervention.

Tracheal extubation time (from discontinuing anesthetics until extubation), Duration of anesthesia (from the injection of anesthetic until discontinuation) duration of the operation (from the injection of anesthetic until until the patient's discharge from the operating room) were recorded for each patient.

We assessed the agitation level with the Pediatric Anesthesia Emergence Delirium (PAED), which provides a score from 0 to 20, at first 15 minutes (T0), 1st (T1), 4th (T4), 8th (T8) and 12th (T12) hours post-extubation

ELIGIBILITY:
Inclusion Criteria:

* patient who will be undergoing adenotonsillectomy with recurrent / chronic tonsillitis or obstructive sleep apnea in the otorhinolaryngology clinic
* American Society of Anesthesiologists (ASA) I-II risk group,
* aged 5-13 years,

Exclusion Criteria:

* patients with history of allergy to any medication used during general anesthesia,
* known or suspected neuromuscular disorders that impair neuromuscular blockade,
* liver and kidney disease,
* asthma,
* bleeding diathesis.
* Written and verbal consents were obtained from the legal guardians of the patients who are blınded of the groups to participate in the study.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Inclusion Criteria:A total of 70 patients in the American Society of Anesthesiologists (ASA) I-II risk group, aged 5-13 years, who will be undergoing adenotonsillectomy
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
agitation level | 1 month
  Pediatric Anesthesia Emergence Delirium (PAED), which provides a score from 0 to 20

SECONDARY OUTCOMES:
pain levels | 1 month
  The pain levels were assessed with visual analogue scale (VAS) scores which assessment scale ranging from 0 to 10 according to the face expression was used

CONTACTS AND LOCATIONS:
Overall Officials: Havva Sayhan, Assis Prof, Study Chair — Sakarya University
Locations (1):
- Sakarya University Research and Training Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mohkamkar M Bs, Farhoudi F Md, Alam-Sahebpour A Md, Mousavi SA Md, Khani S PhD, Shahmohammadi S BSc. Postanesthetic Emergence Agitation in Pediatric Patients under General Anesthesia. Iran J Pediatr. 2014 Apr;24(2):184-90. PMID 25535538